CLINICAL TRIAL: NCT04475549
Title: A Phase 2a Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Individuals With Mitochondrial Encephalomyopathy, Lactic Acidosis, and Stroke-like Episodes (MELAS)
Brief Title: Phase 2a Study of IW-6463 in Adults Diagnosed With Mitochondrial Encephalomyopathy, Lactic Acidosis, and Stroke-like Episodes (MELAS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to enrollment challenges.
Sponsor: Tisento Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C6463-201
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: MELAS
Keywords: mitochondrial disease
MeSH Terms: conditions — MELAS Syndrome; Mitochondrial Diseases

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm study with daily dosing for up to 29 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IW-6463 (Experimental): Open-label IW-6463 15 mg once daily (QD), with possibility to dose reduce to 10 mg.
  Interventions: Drug: IW-6463 Tablets

INTERVENTIONS:
Drug: IW-6463 Tablets — IW-6463 tablets administered orally (daily)
  Other Names: CY6463; zagociguat

SUMMARY:
This is a single-arm study to evaluate safety and tolerability of oral IW-6463 in adults diagnosed with MELAS.

DETAILED DESCRIPTION:
IW-6463 tablets will be orally administered once-daily (QD) for up to 29 days

ELIGIBILITY:
Inclusion Criteria:

1. Prior genetic confirmation of a known mitochondrial disease mutation
2. Neurological features of MELAS (can be based on medical history)
3. Elevated plasma lactate levels at Screening Visit (≥1.0 mmol/L)
4. Women of childbearing potential must have a negative pregnancy test prior to randomization and must agree to use protocol-specified contraception from the Screening Visit through 90 days after the final dose of study drug.
5. Male participants must be surgically sterile by vasectomy (conducted ≥60 days before the Screening Visit or confirmed via sperm analysis) or must agree to use protocol-specified contraception and agree to refrain from sperm donation from the Screening Visit through 90 days after the final dose of study drug.
6. Other inclusion criteria per protocol

Exclusion Criteria:

1. Positive pregnancy test at Screening or on Day 1
2. Hypotension defined as systolic blood pressure (BP) ≤90 mmHg or diastolic BP ≤60 mmHg at Screening or predose at Day 1
3. Hypertension defined as systolic BP >160 mmHg or diastolic BP >100 mmHg, at Screening or predose at Day 1
4. Uncontrolled diabetes
5. Severe gastrointestinal dysmotility as determined by the investigator that may impact compliance and/or oral drug administration, absorption and exposure.
6. Unable to fast for 3-4 hours after a meal
7. Unable or unwilling to adhere to the study schedule, lifestyle restrictions, assessment requirements or, in the clinical judgment of the investigator, is otherwise not suitable for study participation.
8. Current or past history of clinically significant cardiomyopathy and/or cardiac conduction abnormality
9. Used any nicotine-containing products (eg, cigarettes, e-cigarettes, vape pens, cigars) within 1 month of enrollment
10. Other exclusion criteria per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2022-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Glasser, PharmD, Study Director — Cyclerion Therapeutics, Inc.
Locations (5):
- United States (5):
  - Children's National Hospital of DC, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IW-6463
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- IW-6463: Open-label IW-6463 15 mg QD, with possibility to dose reduce to 10 mg.
Arm/Group | IW-6463
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Study Drug Dose Reductions or Discontinuations Due to ≥ 1 Treatment Emergent Adverse Event (TEAE)
Description: A TEAE is defined as an adverse event (AE) with an onset that occurs between the first dose of study drug and the end of study period. AEs are defined as an untoward medical occurrence that does not necessarily have a causal relationship with study drug treatment.
Time Frame: From first dose date to Day 43 (±4)
Measure: Count of Participants; unit: Participants
Arm/Group | IW-6463
Number analyzed (Participants) | 8
Participants
  Dose reduction due to TEAE | 1
  Study drug discontinuation due to TEAE | 0

2. Primary Outcome: Number of Participants Who Experienced ≥1 AE, TEAE, Serious AE (SAE), or TEAE of Special Interest (AESI)
Description: AEs are defined as an untoward medical occurrence that does not necessarily have a causal relationship with study drug treatment. A TEAE is defined as an AE with an onset that occurs from the first dose of study drug up until the end of study period. An SAE is an AE that fulfills 1 or more of the following: results in death; is immediately life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; results in a congenital abnormality or birth defect; is an important medical event that may jeopardize the participant or may require medical intervention to prevent 1 of the outcomes listed above. Events were categorized as mild, moderate, or severe and as related or unrelated to study drug. AESIs include bleeding events, symptomatic hypotensive events and/or tachycardia, dizziness, syncope, and TEAEs related to change of neurobehaviors (ie, suicidality or euphoria).
Time Frame: From first dose date to Day 43 (±4)
Measure: Count of Participants; unit: Participants
Arm/Group | IW-6463
Number analyzed (Participants) | 8
Participants
  Any AE | 8
  Any pretreatment AE | 1
  Any TEAE | 8
  Any severe TEAE | 0
  Any study drug-related TEAE | 4
  Any SAE | 0
  Any TEAE leading to study drug discontinuation | 0
  Any TEAE leading to death | 0
  Any treatment-emergent AESI | 4

ADVERSE EVENTS:
Time Frame: From signing of informed consent (all-cause mortality) or first dose date (adverse events) to Day 43 (±4).
Arm/Group | IW-6463
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IW-6463 (N=8)
Cerebrovascular accident (Nervous system disorders) | 1 — Verbatim term: "metabolic stroke-like event"
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Feeling abnormal (General disorders) | 1
Impaired healing (General disorders) | 1
Oedema peripheral (General disorders) | 2
Blindness transient (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Crystal urine present (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Confusional state (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04475549/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT04475549/SAP_001.pdf